CLINICAL TRIAL: NCT07129902
Title: Contingency Management to Improve Medication for Opioid Use Disorder Continuation After Discharge From the Emergency Department
Brief Title: Contingency Management to Improve Medication for Opioid Use Disorder Continuation After the Emergency Department
Acronym: CM+ED+MOUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Eric A Thrailkill, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5P30GM149331-02 (NIH); 5P30GM149331-02 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: contingency management; medication for opioid use disorder (MOUD); emergency departments; opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): Participants assigned to this arm will receive incentives when they complete their first outpatient MOUD clinic visit and when they complete subsequent visits to pick up their MOUD prescription for the 30-day study period.
  Interventions: Behavioral: Contingency Management; Behavioral: Usual care as prescribed by the ED physicians
- Usual Care (Active Comparator): All participants will receive standard outpatient care at their clinic.
  Interventions: Behavioral: Usual care as prescribed by the ED physicians

INTERVENTIONS:
Behavioral: Contingency Management — Participants in the active arm will receive payment (monetary incentive) contingent on outpatient MOUD treatment attendance.
  Arms: Contingency Management
Behavioral: Usual care as prescribed by the ED physicians — All participants will receive standard outpatient care at their clinic.

SUMMARY:
Project Summary The goal of this pilot clinical trial is to assess contingency management (CM) for increasing attendance at outpatient clinics after Medication for Opioid Use Disorder (MOUD) prescription and clinic referral occurred in the hospital Emergency Department (ED).

* The researchers will compare usual care (UC)+CM to UC alone to see if 1) CM works to promote MOUD clinic attendance after discharge from the ED and 2) demonstrate feasibility of providing CM in the ED and outpatient MOUD clinic settings.
* Researchers will randomize 30 adults who started MOUD in the ED into two conditions. These conditions consist of (A) UC alone: A referral to an outpatient buprenorphine or methadone provider with reminders from STAR program staff or (B) UC+CM: UC plus financial incentives dependent on MOUD clinic attendance to receive an MOUD prescription.

The primary outcome of interest is the number of participants who receive their first MOUD prescription from the outpatient clinic after discharge from the ED in UC+CM compared to the UC-only condition. A secondary outcome will be the proportion of participants who kept attending outpatient MOUD treatment by the end of the 30-day study period between UC+CM and UC conditions. An exploratory outcome will be biochemically-verified illicit opioid abstinence measured at day 30.

DETAILED DESCRIPTION:
Opioid overdose disorder (OUD) and related morbidity and mortality remains an epidemic in the United States with annual deaths surpassing 100,000 in 2021. Medications for Opioid Use Disorder (MOUD) are effective for reducing illicit opioid use and overdose but access to MOUD among US adults with OUD remains low. Hospital Emergency Departments (ED) are a front line in the opioid overdose epidemic. In response to this crisis, a multidisciplinary team in the ED located in the University of Vermont Medical Center (UVMMC) has implemented the Start Treatment and Recovery (STAR) program which consists of dedicated on-site staff in the ED that identify patients with OUD and provide resources, including MOUD prescriptions, and referral to outpatient clinic resources. The STAR program has increased the number of individuals with OUD that enter the ED who receive access to outpatient services and MOUD. Nonetheless, clinic data indicates about 50% of individuals with STAR MOUD referrals attend their first outpatient clinic appointment which highlights a significant gap to be addressed. The present study will use contingency management (CM) to address this gap. CM is a standardized and highly-efficacious treatment that has been applied to reduce opioid use, as well as cigarette, psychostimulant, and alcohol use. The Vermont Center on Behavior and Health has >30 years of experience studying the use of incentives for behavior change. This two-arm pilot randomized clinical trial aims to 1) provide a preliminary test of whether usual care (UC)+CM is more effective than UC alone at promoting MOUD clinic attendance after discharge from the ED and 2) demonstrate feasibility of providing CM in the ED and outpatient MOUD clinic settings. The investigators will randomize 30 adults who initiated MOUD in the ED into two arms. The two arms consist of (A) UC alone: A referral to an outpatient buprenorphine or methadone provider with reminders from STAR program staff or (B) UC+CM: UC plus financial incentives contingent upon MOUD clinic attendance to receive an MOUD prescription. Incentives will be contingent on electronic health records (EHR) indicating a MOUD prescription. Participants will have the opportunity to earn a compensation over 30 days. The incentives will consist of a priming incentive in the ED, a moderate incentive for attending the first outpatient visit, and the remaining incentives distributed evenly according to number of scheduled clinic visits attended. The proportion of participants who receive an MOUD prescription following discharge from the ED is the primary outcome of interest. A secondary outcome will be the proportion of participants who remained in outpatient MOUD treatment at the end of the 30-day study period between UC+CM and UC conditions. An exploratory outcome will be biochemically-verified illicit opioid abstinence measured at day 30. Planned sample size (n=30) is based on previous pilot trials using CM conducted by our group. Although the proposed pilot trial is not powered to detect statistically significant results, the investigators expect effect sizes to be consistent with those found in prior meta-analyses.

ELIGIBILITY:
Major inclusion criteria include

* STAR referral to outpatient clinic (Addiction Treatment Center and Chittenden Clinic) with prescription for buprenorphine or methadone.
* Age ≥18 years.
* Provide informed consent.

Exclusion Criteria

* Pending incarceration in the next 30 days.
* Plan to leave the area (Burlington/Chittenden County) in the next 30 days.
* Physical, health, or structural challenge that prevents attendance at outpatient clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Intake at outpatient MOUD clinic | 30 days
  The proportion of participants who complete their initial (intake) outpatient MOUD clinic appointment after discharge from the emergency department.

SECONDARY OUTCOMES:
Attendance at outpatient MOUD clinic | 30 days
  The proportion of MOUD clinic appointments attended following discharge from the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Thrailkill, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT07129902/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT07129902/ICF_001.pdf